CLINICAL TRIAL: NCT06419673
Title: Induced and Concurrent Serplulimab Plus Chemoradiotherapy Followed by Toripalimab Maintenance Therapy for Stage III-IVA Cervical Cancer: a Prospective, Multicenter, Randomized, Open Controlled Clinical Trial
Brief Title: Serplulimab Plus Chemoradiotherapy for Stage III-IVA Cervical Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, LING YING WU, Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HLX10IIT29
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Cervical Cancer
Keywords: Serplulimab; Concurrent chemoradiotherapy; Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; Carboplatin; Brachytherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serplulimab + chemoradiotherapy , Serplulimab maintenance (Experimental): Participants receive serplulimab 300 mg intravenously (IV) on Day 1 of each 3-week cycle (Q3W) for 3 cycles followed by serplulimab 300 mg IV on Day 1 of each 6-week cycle (Q3W) for an additional 15 cycles. During the Q3W dosing period of serplulimab, participants receive concurrent chemoradiotherapy. The standard of care chemoradiotherapy regimen includes cisplatin 40 mg/m^2 IV or carboplatin (AUC=2) once per week (QW) for 5 or 6 weeks plus external beam radiotherapy followed by brachytherapy not to exceed 8 weeks.
  Interventions: Drug: Serplulimab; Drug: Cisplatin; Drug: Carboplatin; Radiation: Brachytherapy and External Beam Radiotherapy
- Concurrent chemoradiotherapy (Active Comparator): Participants receive concurrent chemoradiotherapy. The standard of care chemoradiotherapy regimen includes cisplatin 40 mg/m^2 IV or carboplatin (AUC=2) once per week (QW) for 5 or 6 weeks plus external beam radiotherapy followed by brachytherapy not to exceed 8 weeks.
  Interventions: Drug: Cisplatin; Drug: Carboplatin; Radiation: Brachytherapy and External Beam Radiotherapy

INTERVENTIONS:
Drug: Serplulimab — Serplulimab will be administered by intravenous infusion at a dose of 300mg on Day 1 of each 21-day cycle until unacceptable toxicity or loss of clinical benefit as determined by the investigator.
  Arms: Serplulimab + chemoradiotherapy , Serplulimab maintenance
Drug: Cisplatin — IV infusion
Drug: Carboplatin — IV infusion
Radiation: Brachytherapy and External Beam Radiotherapy — Brachytherapy and External Beam Radiotherapy

SUMMARY:
This study is a prospective, multicenter, randomized, open controlled clinical trial aimed at evaluating the effectiveness and safety of serplulimab plus chemoradiotherapy in FIGO 2018 stage III or IVA cervical squamous cell carcinoma, adenocarcinoma, and adenosquamous cell carcinoma patients who have not received prior treatment.

DETAILED DESCRIPTION:
Cervical cancer is the most prevalent malignant tumor of the female reproductive system in China, with an estimated 150,700 new cases and 55,700 new deaths annually. Concurrent chemoradiotherapy (CRT) remains the standard treatment for locally advanced cervical cancer (LACC). However, for high-risk LACC (HR-LACC) patients, the 2-year progression-free survival (PFS) rate is only 57%-62%, and the 5-year overall survival (OS) rate is 52%-64%, which are the leading causes of patient mortality. The KEYNOTE-A18 study demonstrated that the combination of pembrolizumab and CRT reduced the progression risk and death risk by 30% and 27%, respectively, for HR-LACC patients. Following this, the FDA approved pembrolizumab in combination with CRT for the treatment of newly diagnosed stages III-IVA cervical cancer in January 2024. This prospective, multicenter, randomized, controlled clinical trial study aims to evaluate the effectiveness and safety of serplulimab induced and combined chemoradiotherapy in FIGO 2018 stage III or IVA cervical squamous cell carcinoma, adenocarcinoma, and adenosquamous cell carcinoma patients who have not received prior treatment.

ELIGIBILITY:
Main Inclusion Criteria:

1. Age ≥ 18 years and ≤ 75 years at time of study entry.
2. Has histologically-confirmed squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma of the cervix.
3. The International Federation of Gynecology and Obstetrics (FIGO) 2018 Stages III-IVA.
4. Diagnosed with PD-L1-positive (combined positive score ≥1).
5. Has not previously received any definitive surgical, radiation, or systemic therapy for cervical cancer.
6. WHO/ECOG performance status of 0 or 1.
7. Patient must have at least one measurable disease as defined by RECIST 1.1.

Main Exclusion Criteria:

1. Has received prior therapy with an anti-programmed cell death receptor 1 (PD-1), anti-programmed cell death receptor ligand 1 (PD-L1), or anti-programmed cell death receptor ligand 2 (PD-L2) agent o..
2. Ongoing participation in another clinical study, or planned initiation of treatment in this study less than 28 days from the end of treatment in the previous clinical study.
3. Known history of serious allergy to any active ingredie or any excipients list in monoclonal antibody.
4. The patient has other factors that, in the judgment of the investigator, may lead to forced early termination of the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival(PFS) at Month 36 | Up to approximately 46 months.
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, or by histopathologic confirmation of suspected disease progression, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. Unequivocal progression of non-target lesions is also considered PD. PFS data will be cumulated to a certain cut-off date and the analysis will be performed via Kaplan-Meier approach to estimate the PFS rate at Month 36 using the entire PFS data up to the cut-off date.

SECONDARY OUTCOMES:
Overall Survival (OS) at Month 36 | Up to approximately 46 months
  Overall Survival (OS) at Month 36 [ Time Frame: Up to approximately 46 months ] OS, defined as the time from initiation of study treatment to death from any cause. OS data will be cumulated to a certain cut-off date and the analysis will be performed via Kaplan-Meier approach to estimate the OS rate at Month 36 using the entire OS data up to the cut-off date. The cut-off date is event-driven and estimated to be approximately 46 months.
Objective Response Rate (ORR) | Baseline up to approximately 36 months
  ORR is defined as the percentage of participants who have a Complete Response (CR: Disappearance of all target and non-target lesions and also includes reduction of all nodal lesions to <10mm) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions and includes no unequivocal progression in non-target lesions) per RECIST 1.1.
Complete Response Rate（CRR） | Baseline up to approximately 36 months
  The rate of CR (Disappearance of all target and non-target lesions and also includes reduction of all nodal lesions to <10mm).
Time to the first disease progression （TTP） | Up to approximately 24 months
  Ddefined as the interval between the date of the initial medication and the time of imaging progression.
Duration of response (DOR) | Up to approximately 24 months
  Duration of response is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: LINGYING WU, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China